CLINICAL TRIAL: NCT02105259
Title: Internet-delivered Psychodynamic Therapy for Social Anxiety Disorder: A Randomized Controlled Trial
Brief Title: Internet-delivered Psychodynamic Therapy for Social Anxiety Disorder (SOFIA)
Acronym: SOFIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Karolinska Institutet (Other); Stockholm University (Other)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GA-ANX2014-APT
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Last update posted 2023-10-05 (Actual); Status verified 2015-08

CONDITIONS: Social Anxiety Disorder
Keywords: Test; psychodynamic; Internet-delivered psychodynamic treatment; patients with social anxiety disorder
MeSH Terms: conditions — Phobia, Social | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Psychodynamic Internet Treatment (Experimental): Psychodynamic Internet Treatment for social anxiety disorder during 10 weeks and guided by a psychologist
  Interventions: Behavioral: Psychodynamic Internet Treatment
- Waiting list with support (Active Comparator): Behavioral: supportive check-ups via the Internet during 10 weeks
  Interventions: Other: Waiting list

INTERVENTIONS:
Behavioral: Psychodynamic Internet Treatment — Psychodynamic Internet Treatment for patients social anxiety disorder
  Arms: Psychodynamic Internet Treatment
Other: Waiting list — Waiting list, where participants wait for delayed treatment
  Arms: Waiting list with support

SUMMARY:
The overall aim of this study is to develop and test a psychodynamic Internet--delivered psychological treatment for patients with social anxiety disorder and compare its efficacy to a waiting list.

DETAILED DESCRIPTION:
Participants with social anxiety disorder (MINI telephone interview) will be recruited via mass media and randomly allocated to psychodynamic Internet--delivered psychological treatment or to a waiting list control condition.

ELIGIBILITY:
Inclusion Criteria:

* Social anxiety disorder as diagnosed by the MINI diagnostic interview

Exclusion Criteria:

* Severe depression

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Liebowitz Social Anxiety Scale | Baseline and End of treatment (10 weeks)

SECONDARY OUTCOMES:
Patient Health Questionnaire Depression 9 item | Baseline
Patient Health Questionnaire Depression 9 item | End of treatment (10 weeks)
Patient Health Questionnaire Anxiety 7 item | Baseline
Patient Health Questionnaire Anxiety 7 item | End of treatment (10 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, Principal Investigator — Linkoeping University
Locations (1):
- Department of Behavioural Sciences and Learning, Linköping University, Linköping, Sweden

REFERENCES:
- [Derived] Johansson R, Hesslow T, Ljotsson B, Jansson A, Jonsson L, Fardig S, Karlsson J, Hesser H, Frederick RJ, Lilliengren P, Carlbring P, Andersson G. Internet-based affect-focused psychodynamic therapy for social anxiety disorder: A randomized controlled trial with 2-year follow-up. Psychotherapy (Chic). 2017 Dec;54(4):351-360. doi: 10.1037/pst0000147. PMID 29251954